CLINICAL TRIAL: NCT05803278
Title: Application of an Online Screening and Empowerment Program Carried Out at Schools to Identify Children With Specific Learning Disorders
Brief Title: Online Screening and Empowerment Program for Children With SLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC 23/20
Record Dates: First submitted 2023-03-24; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Learning Disorder
Keywords: Specific Learning Disorders; Screening; Online enhancement
MeSH Terms: conditions — Learning Disabilities; Specific Learning Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children positive to screening test (Experimental): Children positive to the online test "InTempo", which includes standardized and scientifically validated tests in the following areas: Metaphonology, Reading and Writing
  Interventions: Other: Online enhancement training

INTERVENTIONS:
Other: Online enhancement training — Online enhancement training lasting 3 months, using the "InTempo" app system (Gea-Metaphonology-Athena-reading/Ermes-writing) three times a week for twenty minutes. The training will include: Metaphonological Enhancement; Reading Enhancement; Writing Enhancement.

SUMMARY:
One of the problems faced by health services that deals with the diagnosis and treatment of Specific Learning Disorders (SLD), like Dyslexia, Dysgraphia, Dysorthography and Dyscalculia, is the long waiting lists for first visits to possible confirm the diagnosis. One of the reasons explaining the long waiting times is that the school refers a large number of children to the hospital services who do not actually have SLD but a simple school difficulty. These two are very different conditions:

* SLD is a neurobiological and genetic-based disorder that, with various degrees of severity, lasts a lifetime. Epidemiological data of the FVG region report a prevalence of dyslexia of 3.1%. Therefore, a prevalence of SLD between 4 and 5% can be assumed. This is a condition whose expressiveness cannot be modified by an enhancement intervention;
* The school difficulties are not innate and are characterized by an initial slowdown in bed-writing learning. The prevalence of low-performance school difficulties is between 10 and 15%. This type of problem improves significantly following specific enhancement.

Resistance to enhancement intervention is precisely one of the criteria that is still used to distinguish a school difficulty from a SLD: students with SLD would be those who show resistance to specific educational interventions. This criterion is based on the assumption that SLD has a precise neurofunctional basis in contrast to school difficulties. These are a transitional condition, which can be modified by didactic adaptations and enhancement activities (Law 170/2010; regional resolution 933/2014 FVG).

The application of enhancement tools in the school environment would therefore make it possible to distinguish, on the basis of the response, subjects with simple school difficulties from those with suspected SLD and, therefore, to report just those one, to the health services for diagnostic confirmation, contributing to the reduction of the workload of the hospital services and the reduction of waiting lists. These results are very important for children with SLD who could be identified and treated in an early and timely manner. The aim of this project is to apply an online screening and further school enhancement process using the "InTempo software" to distinguish children with SLD from those with school difficulties, thus also obtaining data on the real incidence of SLD and school difficulties in The Friuli Venezia Giulia Region.

ELIGIBILITY:
Inclusion Criteria:

* Children attending the second year of the primary school (about 7-8 years of age)

Exclusion Criteria:

* Presence of biological problems associated to school difficulties
* Low cognitive level

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1548 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Prevalence of SLD | 6 months
  The first screening test and the subsequent enhancement training for positive will be carried out on-line in school children aged 7-8 years. Children without improvement after enhancement training (second screening test) will be considered positive (presence of SLD) and sent to the health services for a specific diagnostic evaluation.

SECONDARY OUTCOMES:
To evaluate the prevalence of school difficulties | 6 months
  Defined by positivity at the first screening test and by negativity at the second, carried out after the enhancement intervention
To compare the Strengths and Difficulties Questionnaire scores recorded during the study | 6 months
  The Strengths and Difficulties Questionnaire (italian version) will be administered to parents of the children involved in the study pre and post intervention to evaluate emotional and behavioural characteristics of the children and to assess how they change during the enhancement process.

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Lonciari, MSC, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided